CLINICAL TRIAL: NCT05306938
Title: Adolescent Wellness Visits in Tanzania
Acronym: VITAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other); Duke University (Other); Arizona State University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 21-1198; 5R01HD102279 (NIH)
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: HIV Testing; Contraceptive Usage
Keywords: HIV testing and counseling; Adolescent health; Mental health; Contraception
MeSH Terms: conditions — Contraception Behavior; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This is a cluster randomized control trial, with randomization occurring at the school level into one of two arms: intervention or control.
Who Masked: Outcomes Assessor
Masking Description: Statisticians will be blinded to the intervention status of individuals and schools.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Adolescents in this arm will receive the Adolescent Wellness Visit intervention.
  Interventions: Behavioral: Adolescent Wellness Visit
- Control (No Intervention): Adolescents in this arm will not receive the Adolescent Wellness Visit intervention.

INTERVENTIONS:
Behavioral: Adolescent Wellness Visit — Adolescent Wellness Visits (AWVs) are a new health service platform for reaching young adolescents with HTC and other evidence-based prevention services which are clinic-based and school-facilitated. The AWVs bundle the following health screenings, education, and counseling on: nutrition, vision, dental, mental health (depression), contraception, sexually transmitted infections, and optional HIV testing.
  Arms: Intervention

SUMMARY:
This study evaluates the impact of clinic-based 'Adolescent Wellness Visits' (AWVs) coordinated with primary schools that offer a package of evidence-based adolescent-friendly preventative services on HIV testing uptake in Tanzania.

Participants: The clinical trial participants are approximately 1500 adolescents in their final year of primary school who will be enrolled in this cluster randomized controlled trial (RCT) from 20 primary schools and followed up for two years post-primary school.

[Qualitative data from approximately 250 adult stakeholders will also be collected via focus group discussions (FGDs) and in-depth interviews (IDIs) for implementation science, non-trial related study aims] .

Procedures: Adolescent data will include surveys with self-report measures and reviews of their medical records (using REDCap). The adult qualitative data will be in the form of translated and transcribed FGD and IDI transcripts as Word documents.

DETAILED DESCRIPTION:
In most low-resource country settings, there is no routine clinic-based adolescent health check-up after the recommended child wellness visits end at age 5. Adolescents in low-resource settings need a preventative health service platform applicable for all young people that promotes a culture of health-seeking behavior. This study evaluates the impact of Adolescent Wellness Visits (AWVs), a new health service platform, for reaching young adolescents with HIV testing and counseling (HTC) and other evidence-based prevention services which are clinic-based and school-facilitated. AWVs could meet the reproductive health needs of at-risk adolescents and have a larger public health impact for all adolescents on access to traditionally neglected and under-treated health conditions such as poor nutrition, and vision, dental, and mental health problems at the time of delivery as well as in the future as adolescents continue with more timely service utilization.

The AWV is designed to be delivered during the last year of primary school when school attendance is high, and adolescents are on the cusp of puberty (mean age 13). This project is a collaboration between the University of North Carolina at Chapel Hill in the United States (prime), Muhimbili University of Health and Allied Sciences in Dar es Salaam, Tanzania, and Duke University in the United States.

Specific Aims are:

1. To assess the impact of Adolescent Wellness Visits on HTC (for all adolescents; primary outcome) and contraceptive uptake (for a sexually active subset) up to two years post-primary school via a cluster randomized controlled trial (20 school-clinic pairs: 10 intervention + 10 control; n= approximately 1500 adolescents);
2. To evaluate factors that support or limit implementation of the AWV model and fidelity/adherence to implementation of the proposed package of evidence-based practices included in the AWV by utilizing 24 focus group discussions (FGDs) with implementers and 60 semi-structured interviews (IDIs) with key informants; and
3. To evaluate the cost-effectiveness of AWVs on two key health behavioral outcomes: uptake of HTC for all adolescents, and reductions in unmet need for contraception among sexually active adolescents.

Methodology:

Participants: Up to 1,500 adolescents in the seventh and final grade of primary school; about 650 for each randomized study arm (10 intervention schools + 10 control schools).

Study design: Investigators will implement this cluster RCT with 10 intervention schools and 10 control schools. Randomization occurs at the school level and both adolescent assent and parental consent will be obtained for all participants. There are 4 data collection timepoints (baseline, follow-up 1, follow-up 2, follow-up 3/endline). At baseline, for control schools, adolescents will be interviewed at their schools or in the community while for intervention schools, adolescents will be interviewed before and after their AWV at the clinic. The AWV intervention will involve a single adolescent wellness visit to a public health facility within a walking distance (1 Km) that offers a package of government-approved, evidence-based youth-friendly services (screenings for nutrition, vision, dental pain, mental health, puberty and contraception information and counseling, syndromic sexually transmitted infection screening, and optional HIV testing) in Dar es Salaam and Pwani regions in Tanzania. All children (intervention and control) will be given a Tanzanian government endorsed Puberty Book and encouraged to ask questions to teachers/parents and guardians (intervention participants will also have the opportunity to ask questions with clinical staff during AWV). Follow-interviews with adolescents will be community-based.

Direct observations coupled with FGDs and IDIs (perspectives of parents, direct providers of health and education services and other key stakeholders), will describe factors that support or limit implementation of the AWV model including fidelity/adherence to components of the evidence-based package.

ELIGIBILITY:
Inclusion Criteria:

* At enrollment, must be a student in the seventh and final year of primary school.

Exclusion Criteria:

* Youth that are out of school at the time of enrollment.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1095 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Proportion of adolescents who self-reported HIV testing and counseling over 24-month follow-up, inclusive of the Adolescent Wellness Visit | Approximately 24 months, inclusive of AWV.
  Data will be collected at four time points via individual interviews between the adolescent and a research assistant at the AWV (baseline), and at follow-up 1, follow-up 2, and follow-up 3/endline. At each time point, the adolescent will be asked whether they have had an HIV test since the previous interview. The AWV intervention is delivered concurrently with baseline data collection.
Proportion of adolescents who self-reported HIV testing and counseling over 24-months follow-up, exclusive of the Adolescent Wellness Visit | Approximately 24 months, excluding AWV.
  Data will be collected at four time points via individual interviews between the adolescent and a research assistant at the AWV (baseline), and at follow-up 1, follow-up 2, and follow-up 3/endline. At each time point, the adolescent will be asked whether they have had an HIV test since the previous interview. The AWV intervention is delivered concurrently with baseline data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Joy Noel Baumgartner, PhD, MSSW, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared per NIH requirements in the public repository and no later than 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol, SAP
Time Frame: 9 to 36 months following publication or per NIH requirements
Access Criteria: Investigator proposing to use the data has IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC or publicly available via NIH repository.

REFERENCES:
- [Derived] Alexander K, Gitagno D, Mtei RJ, Minja A, Lema I, Egger JR, Van Praag E, Kaaya S, Baumgartner JN. Caregiver attitudes towards HIV testing and contraceptive services for adolescents in Tanzania. AIDS Care. 2026 Jan;38(1):83-96. doi: 10.1080/09540121.2025.2569975. Epub 2025 Oct 15. PMID 41093752

DOCUMENTS (1):
  • Informed Consent Form (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT05306938/ICF_000.pdf